CLINICAL TRIAL: NCT02937597
Title: The Effect of an E-learning Proficiency Based Progression Training Programme for Clinical Communication on ISBAR Performance
Brief Title: E-learning Proficiency Based Progression Training Programme for Clinical Communication on ISBAR Performance (eISBAR)
Acronym: eISBAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Nora McCarthy, Lecturer in Medical Education, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: eISBAR
Record Dates: First submitted 2016-10-16; First posted 2016-10-18 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Communication
Keywords: proficiency based progression; feedback; computer based assessment; non technical skills; deteriorating patient; ISBAR
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- National e-learning programme only (HSE) (Active Comparator): Active Comparator: National e-learning programme only (HSE) National e-learning programme only Recent successful completion of the National e-learning programme by certificate will be displayed. Students then undergo performance assessment via low fidelity simulation and complete a questionnaire.
  Interventions: Behavioral: HSE
- eS: eScenarios (Active Comparator): Recent successful completion of the National e-learning e-learning programme by certificate will be displayed. Students will proceed to an online learning course with 4 scenarios to work through but no requirement to meet a proficiency benchmark. Following training students undergo performance assessment via low fidelity simulation and complete a questionnaire.
  Interventions: Behavioral: eS: eScenarios
- ePBP: eProficiency Based Progression (Experimental): Recent successful completion of the National e-learning programme by certificate will be displayed. Students will proceed to a PBP e-learning course using the same series of cases as S. PBP students will be scored according to predefined metrics and will be required to reach proficiency benchmarks for the cases within the e-learning course to allow progression through the cases. Following training students undergo performance assessment via low fidelity simulation and complete a questionnaire.
  Interventions: Behavioral: ePBP: eProficiency Based Progression

INTERVENTIONS:
Behavioral: ePBP: eProficiency Based Progression — National e-learning programme plus Proficiency-based progression through 4 scenarios in an online learning course and facilitator when requested
  Arms: ePBP: eProficiency Based Progression
Behavioral: eS: eScenarios — National e-learning programme plus access to 4 scenarios in an online learning course and facilitator when requested
  Arms: eS: eScenarios
Behavioral: HSE — National HSE e-learning programme only
  Arms: National e-learning programme only (HSE)

SUMMARY:
Objective:

To determine the effectiveness of proficiency based inter-professional communication training in an online environment on medical student's use of the ISBAR (Identify, Situation, Background, Assessment, Recommendation) communication escalation protocol in the deteriorating patient

Setting: The study will be conducted in University College Cork, Ireland. Participants: Fifth year medical students, who are scheduled to undertake ISBAR training as part of the National Early Warning Score (NEWS) programme.

Intervention: Participants will be prospectively randomized to one of three groups for training before undertaking a performance assessment of an ISBAR communication relevant to a deteriorating patient in a low fidelity simulation environment: HSE group (the national e-learning programme only); S group (national e- learning plus access to online scenarios and facilitator when requested) and PBP group (national e-learning plus access to online scenarios training course with in-built proficiency-based progression, and facilitator when requested).

Main outcome and measures: A proficiency benchmark on the performance of ISBAR communication in the context of an acutely deteriorating patient.

DETAILED DESCRIPTION:
The first successful simulation validation study used a proficiency-based progression methodology. Since then the approach has been successfully deployed to produce superior technical skills but has not yet been validated for non-technical (communication) skills. It has also not yet been validated through the medium of virtual learning. The ISBAR (Identify, Situation, Background, Assessment and Recommendation) has been selected as the standardised tool for clinical communication in relation to an acutely deteriorating patient in many healthcare organisations worldwide, including Ireland.

The aim of this study is to explore whether proficiency-based progression (PBP) could be applied to an e-learning training course for ISBAR performance to produce a superior skill set.

The study will compare performance outcomes of students who receive the national e-learning programme only with those who receive it in combination with either standard e-learning course with scenarios or proficiency-based progression (PBP) e-learning course with scenarios.

Participants will be prospectively randomized to one of three training groups. Following a pre-test observation through low-fidelity simulation, they will then undergo their respective training courses before undertaking a post-test performance assessment of an ISBAR communication relevant to a deteriorating patient in a low fidelity simulation environment:

1. Online learning only (HSE) -the national e-learning programme only
2. Scenarios (S) -national online learning plus online scenario course training
3. Proficiency based progression (PBP) -national online learning plus proficiency-based progression online scenario course training.

Main outcome and measures: A proficiency benchmark on the performance of ISBAR communication in the context of an acutely deteriorating patient.

All participants will be required to supply baseline demographic information before undertaking the training.

Performance metrics have previously been identified, operationally defined and agreed upon at a modified Delphi panel meeting consisting of medical experts for a series of paper-based simulation cases and a standardised high fidelity simulation case used as the assessment case. This case will be used in this study in a low fidelity environment. The proficiency benchmark for each case has been set based on the performance of experienced medical personnel on each case as a series of steps, errors and critical errors.

Outcome assessment will be scored by reviewing auditory recordings of ISBAR performance by each participant on the standardised case in the low fidelity simulated environment.

ELIGIBILITY:
Inclusion Criteria:

* final year medical students in UCC

Exclusion Criteria:

* lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-10; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Proportion of those reaching the benchmark on the assessment case | 12 months
  Independent review by two blinded assessors of audio recorded ISBAR phone call conducted in the low fidelity simulation setting

SECONDARY OUTCOMES:
recording of data in learning management system for various course attempts | 12 months
  recording of data in learning management system for various course attempts
Number of completed steps | 12 months
  Number of successfully completed steps as predefined by the metrics for the assessment case

OTHER OUTCOMES:
Number of total errors | 12 months
  Number of total errors as predefined by the metrics for the assessment case
Number of errors/critical errors | 12 months
  Number of errors/critical errors as predefined by the metrics for the assessment case
Number of attempts required to reach proficiency on each of the 4 cases in ePBP | 12 months
  Number of attempts required to reach proficiency on each of the 4 cases as recorded by the e-learning course ePBP

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Gallagher, PhD, Study Director — Director Technology Enhanced Learning ASSERT, UCC
Locations (1):
- University College Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallagher AG, Seymour NE, Jordan-Black JA, Bunting BP, McGlade K, Satava RM. Prospective, randomized assessment of transfer of training (ToT) and transfer effectiveness ratio (TER) of virtual reality simulation training for laparoscopic skill acquisition. Ann Surg. 2013 Jun;257(6):1025-31. doi: 10.1097/SLA.0b013e318284f658. PMID 23426342
- [Background] Angelo RL, Ryu RK, Pedowitz RA, Beach W, Burns J, Dodds J, Field L, Getelman M, Hobgood R, McIntyre L, Gallagher AG. A Proficiency-Based Progression Training Curriculum Coupled With a Model Simulator Results in the Acquisition of a Superior Arthroscopic Bankart Skill Set. Arthroscopy. 2015 Oct;31(10):1854-71. doi: 10.1016/j.arthro.2015.07.001. Epub 2015 Sep 2. PMID 26341047
- [Background] Van Sickle KR, Ritter EM, Baghai M, Goldenberg AE, Huang IP, Gallagher AG, Smith CD. Prospective, randomized, double-blind trial of curriculum-based training for intracorporeal suturing and knot tying. J Am Coll Surg. 2008 Oct;207(4):560-8. doi: 10.1016/j.jamcollsurg.2008.05.007. Epub 2008 Jul 14. PMID 18926460
- [Derived] McCarthy N, Neville K, Pope A, Barry L, Livingstone V. Effectiveness of a proficiency-based progression e-learning approach to training in communication in the context of clinically deteriorating patients: a multi-arm randomised controlled trial. BMJ Open. 2023 Aug 3;13(8):e072488. doi: 10.1136/bmjopen-2023-072488. PMID 37536965